CLINICAL TRIAL: NCT02790684
Title: A Study Assessing the Mass Balance of a Single Oral Dose of [14C] DS-8500a in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DS8500-A-U112
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2017-09

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — firuglipel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DS-8500a (Experimental)
  Interventions: Drug: DS-8500a

INTERVENTIONS:
Drug: DS-8500a

SUMMARY:
This is a Phase 1, open-label, single-center, non-randomized study to assess the mass balance of a single oral dose of DS-8500a in healthy male subjects, 18 years (y) to 60 y of age, inclusive. The radiolabeled investigational medicinal product will be administered to 12 healthy male subjects in 2 cohorts of 6 subjects each.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 years (y) and 60 y of age, inclusive.
* Subjects must have a body mass index (BMI) of 19 kg/m2 to 30 kg/m2, inclusive; or, if outside the range, not clinically significant and agreed with Sponsor and primary investigator (PI).
* Subjects must be in good health as determined at Screening and Day -1 (Check-in) assessed by medical history (Screening only), physical examination, vital signs, hematology, virology (Screening only), and urinalysis.
* Laboratory results (serum chemistry, hematology, and urinalysis) must not be outside the normal range or if outside the normal range, then the PI considers the value not clinically relevant.
* Subjects must agree not to participate in any other investigational study until the end of the trial.
* Subjects must be willing to abstain from grapefruit/grapefruit juice and Seville oranges from 10 d before the first dose of study medication and throughout the study.
* Subjects must be willing to refrain from consuming food or beverages containing caffeine/xanthine and alcohol starting 24 h prior to Check-in on Day -1.
* Subjects must be able to understand and willing to comply with all study requirements, and willing to allow the collection of all blood, fecal, and urine specimens.
* Subjects must give written informed consent to participate in the study prior to Screening. Consent will be documented by the subject's dated signature that will be counter signed and dated by a witness. The appropriate HIPAA authorization forms must be signed and dated by the subject.
* Male subjects must agree to contraception (condom with spermicide) in addition to having their female partner (if of childbearing potential) use another form of contraception (eg, an intrauterine device, diaphragm with spermicide, oral contraceptive, injectables, or subdermal hormonal implant) from the first dose until 12 wk following the last dose administration. Also, male subjects must not donate sperm for a period of 12 wk following drug administration.
* Subject must have a history of regular bowel movements (defined in this instance as a bowel movement at least every other d without the need for medication).
* Subjects must be willing to eat entire meals and snacks provided during the stay at the research facility and understand that the diet will include foods with high fiber content and possibly prune juice.

Exclusion Criteria:

* Subjects who have received any prescription or non-prescription (over-the-counter [OTC]) systemic medication, topical medication, or herbal supplement (including St. John's Wort [hypericin]) within 14 d prior to dosing.
* Subjects who participated in a clinical study involving administration of an investigational drug (new chemical entity), or a marketed drug within 30 d or 5 half-lives of that investigational drug or marketed drug prior to dosing.
* Subjects who were administered radiolabeled substances or exposed to significant radiation (eg, serial X-rays or computed tomography (CT) scans, barium meal, occupational exposure etc) within 12-mo of dosing.
* Subjects who have been involved in an occupation that requires monitoring for radiation exposure (eg, X-ray technician).
* Liver function (aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin [TBL]) test results range should not be be > upper limit of normal at Screening and during Enrollment on Day -1.
* Subjects with an estimated glomerular filtration rate (eGFR) (using Modification of Diet in Renal Disease [MDRD] equation) < 90 mL/min.
* Subjects with Fridericia's corrected QT interval (QTcF) interval duration > 450 ms, obtained as an average from the 3 ECG recorder's measurements on triplicate Screening ECGs (3 ECGs in close succession at least 1 min apart) taken after at least 10 min of quiet rest in the supine position.
* Subjects with abnormal waveform morphology on any of the ECGs at the Screening and on Day -1 that would preclude accurate measurement of the time for both ventricular depolarization and repolarization (QT) interval duration.
* Subject who have participated in a previous DS-8500a study within 6-mo prior to the screening.
* Subjects with a history of significant allergic response to any drug except penicillin.
* Subjects with a history of any serious disorder, including cardiovascular, hematologic, pulmonary, hepatic, renal, gastrointestinal, connective tissue disease, uncontrolled endocrine/metabolic, oncologic (within the last 5 y), neurologic, and psychiatric diseases, or any disorder that may prevent the successful completion of the study.
* Subjects who consume more than 28 units of alcohol per wk (one unit of alcohol equals one-half pint of beer, 4 oz of wine, or 1 oz of spirits) or those subjects who have a significant history of alcoholism or drug/chemical abuse within 2 y prior to Screening.
* Subjects who have used tobacco products or nicotine-containing products (including smoking cessation aids, such as gums or patches) within 6-mo prior to dosing.
* Subjects with positive results on tests for drugs of abuse, cotinine, or alcohol at Screening and on Day -1.
* Subjects who test positive for HBsAg, or antibody to HCV or HIV, at Screening.
* Subject is employed by the clinic.
* Subjects who have a familial relationship with another study participant.
* Subjects who, in the opinion of the PI, should not participate in the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
total 14C radioactivity in urine and feces | Day 1 to Day 21
  to determine mass balance (excretion) of DS-8500a

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of DS-8500a | Day 1 to Day 21
  determine the pharmacokinetics of DS-8500a
Time of maximum concentration (Tmax) of DS-8500a | Day 1 to Day 21
  determine the pharmacokinetics of DS-8500a
Area under the concentration curve (AUC) of DS-8500a | Day 1 to Day 21
  determine the pharmacokinetics of DS-8500a
number and severity of adverse events | Day 1 to Day 21
  to determine the safety and tolerability of DS-8500a

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/